CLINICAL TRIAL: NCT03326635
Title: Prevalence Study : Elderly Patients and Rehabilitation in ICU. Impact of Frailty.
Acronym: FRAGIREA
Status: Completed | Type: Observational
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 69HCL17_0017
Record Dates: First submitted 2017-10-17; First posted 2017-10-31 (Actual); Last update posted 2019-08-14 (Actual); Status verified 2019-08

CONDITIONS: Resuscitation
Keywords: Resuscitation; Frailty; ICU; Ageing; Rehabilitation; Elderly
MeSH Terms: conditions — Frailty | interventions — Aging; Intensive Care Units

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- frailty group: frailty score ≤ 3
  Interventions: Other: Frailty in elderly (≥70 y) patients in ICU
- non-frailty group: frailty score >3
  Interventions: Other: Frailty in elderly (≥70 y) patients in ICU

INTERVENTIONS:
Other: Frailty in elderly (≥70 y) patients in ICU — Determine the prevalence of frailty in elderly patients (≥ 70 year old) in a group of French ICUs. The frailty is measured by a score (Fried score) at the admission of the patient

SUMMARY:
Study design. The study FRAGIREA is a multicentric prevalence study on the frequency of frailty among elderly patients and the quality of management. The voluntary ICUs will have to include all patients ≥ 70 years on a limited period (1 month) or until the number of 15 inclusions is reached. The frailty is going to be evaluated by a frailty score adapted to the ICU, based on informations given by the patient's family.

It is a descriptive non-interventional study, aiming at the description of frequency of frailty and management of the patient in order to set-up a prospective future study on the potential role of early rehabilitation of ageing patients in ICUs.

ELIGIBILITY:
Inclusion Criteria:

* ≥ 70 year-old
* Prevision of a length of stay > 24 hrs.
* Patient or relative who received information about the study and did not oppose it

Exclusion Criteria:

* Life expectancy < 24 hrs
* Patients unable to communicate and no next of kin available.
* adults, non-emancipated minors, persons unable to receive information,
* persons placed under the safeguard of justice,
* subject participating in another search including an exclusion period still in progress at pre-inclusion

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Patients ≥ 70 year-old admitted to an ICU.
Sampling Method: Non-Probability Sample
Enrollment: 527 (Actual)
Dates: Start 2018-04-08 (Actual); Primary Completion 2019-01-25 (Actual); Study Completion 2019-07-24 (Actual)

PRIMARY OUTCOMES:
Frailty in elderly (≥70 years old) patients in intensive care unit (ICU) | One month or 15 patients ≥ 70 years old
  We assessed the 5 components of Fried's frailty index, resulting from cumulative decline across multiple physiological systems and contain five criteria (shrinking, weakness, slowness, low-level physical activity, and self-reported exhaustion). All five components were considered from the previously reported definition and adapted to the ICU environment. The patients were considered to be frail if they had three or more frailty components among the five criteria.

SECONDARY OUTCOMES:
Organ failures | About 8 days
  During the patients' hospitalization in ICU, the following data were collected last day in ICU:
  the need for dialysis during ICU the duration of mechanical ventilation (number of days under mechanical ventilation) the duration of shock (number of days under catecholamines)
Nutritional support | About 8 days
  Nutritional intake during ICU stay, from the first day to the patient's exit, including route of administration (enteral, parenteral), last day in ICU we assessed:
  number of days under enteral nutrition number of days under enteral parenteral nutrition calculation of the average calorie / day
Rehabilitation | About 8 days
  Last day in ICU, we record the highest level of mobilization achieved during the ICU period, the following ordinal scale was used: 1) no mobilization, 2) turning in bed, 3) sitting in bed with the head of bed elevated, 4) sitting on the edge of the bed with feet on floor, 5) sitting out of bed in a chair, 6) standing out of bed, 7) marching in place, 8) walking, 9) using cycloergometer and 9) using electrical muscle stimulation.
Mortality | 90 days
  ICU mortality and Hospital mortality Decision of therapeutics limitation. Length of stay (ICU and hospital stay).

CONTACTS AND LOCATIONS:
Locations (37):
- France (36):
  - CH Aix en Provence, Aix-en-Provence
  - CHU Angers, Angers
  - CH Annecy, Annecy
  - CH Annonay, Annonay
  - CH Argentueil, Argenteuil
  - CH Belfort, Belfort
  - CH Béziers, Béziers
  - CH Bourg en Bresse, Bourg-en-Bresse
  - CH Bourgoin-Jallieu, Bourgoin
  - CH Chalons sur Saône, Chalon-sur-Saône
  - CH Chambéry, Chambéry
  - CHU Clermont-Ferrand, Clermont-Ferrand
  - CH Sud Francilien, Évry
  - CHU Grenoble, La Tronche
  - Hôpital Edouard Herriot, G Réa, Lyon
  - Hôpital Edouard Herriot, N réa, Lyon
  - Hôpital Edouard Herriot, P Réa, Lyon
  - Hôpital de la Croix Rousse, Lyon
  - AP-HM Hôpital Nord, Marseille
  - AP-HM La Timone, Marseille
  - CH Montauban, Montauban
  - CH Montélimar, Montélimar
  - CH Moulins, Moulins
  - CHU Nantes, Nantes
  - CHU Nice, Nice
  - Centre Hospitalier Lyon Sud Réa Nord, Pierre-Bénite
  - Centre Hospitalier Lyon Sud, Pierre-Bénite
  - CHU Poitiers, Poitiers
  - CHU de Rennes, Rennes
  - CHU Rennes, Rennes
  - CHU Rouen, Rouen
  - CH Saint Denis, Saint-Denis
  - CHU Hôpital Nord, Saint-Etienne
  - CH Salons de Provence, Salon-de-Provence
  - CH Valence, Valence
  - CH Vichy, Vichy
- CH Mayotte, Mayotte, Mayotte